CLINICAL TRIAL: NCT05947292
Title: PLEXUS (Pediatric Lower Extremity Ultrasound-Guided Nerve Block) Study: A Prospective, Multi-center, Observational Study Comparing Ultrasound Guided Fascia Iliaca Compartment Nerve Block to Systemic Analgesia for Femur Fractures in the Pediatric Emergency Department
Brief Title: Study Comparing Ultrasound-guided FICNB Block to Systemic Analgesia in Treatment of Pediatric Femur Fracture
Acronym: PLEXUS
Status: Completed | Type: Observational
Sponsor: Zachary Binder (Other)
Collaborators: University of Michigan (Other); Medical University of South Carolina (Other); Yale University (Other); Emory University (Other); University of California, San Diego (Other); University of California, San Francisco (Other); Denver Health and Hospital Authority (Other); Children's Hospital of The King's Daughters (Other); Gold Coast Hospital and Health Service (Other Government)
Responsible Party: Sponsor-Investigator, Zachary Binder, Assistant Professor, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: STUDY00000295
Record Dates: First submitted 2023-06-14; First posted 2023-07-17 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nerve Block: Patients with femur fractures who receive a fascia-iliaca compartment nerve block as part of their care in the Emergency Department.
  Interventions: Procedure: Ultrasound-Guided Fascia Iliaca Compartment Nerve Block
- No Nerve Block: Patients with femur fractures who receive only intravenous analgesia in the Emergency Department.

INTERVENTIONS:
Procedure: Ultrasound-Guided Fascia Iliaca Compartment Nerve Block — Patient's who receive this intervention will have an ultrasound-guided fascia iliaca compartment nerve block performed in the Emergency Department.
  Groups: Nerve Block

SUMMARY:
The goal of this prospective observational study is to compare pain control strategies in children with femur fractures. Researchers will compare ultrasound-guided fascia iliaca compartment nerve block to IV pain control alone. The main questions it aims to answer are:

* Are ultrasound-guided fascia iliaca compartment nerve blocks as effective as IV pain control in controlling pain?
* Do patients who receive an ultrasound-guided fascia iliaca compartment nerve block require less opioid pain medication than those that don't?

Participants will be asked to provide pain scores during their Emergency Department stay. Participants parents will be asked to complete a brief survey at the time their child is leaving the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* Acute femur fracture (less than 24 hours from initial injury)
* Glasgow Coma Scale of 14 or greater at time of enrollment

Exclusion Criteria:

* Allergy or hypersensitivity to local anesthetic agents
* Pregnant
* Prisoner
* Neurovascular injury to the affected limb
* Bilateral femur fractures
* Confirmed, or significant clinical suspicion for, injury to their head, neck, chest, abdomen, back or pelvis
* Imaging suggestive of a head, neck, chest, abdomen, back or pelvic injury
* Laboratory results suggestive of a head, neck, chest, abdomen, back or pelvic injury
* A fracture not limited to the extremities (i.e. vertebral compression fracture)
* A significantly displaced extremity fractures (aside from the primary femur fracture)
* An open fracture (aside from the primary femur fracture)
* An additional fracture to the limb of the primary femur fracture (i.e. tibia fracture in the same leg as the primary femur fracture).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 4-18 hears of age who present to the Emergency Department with an acute isolated femur fracture.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
60 Minute Pain Score | 60 minutes after enrollment.
  Self reported pain score using the Faces Pain Scale-Revised. Values range from 1-10 (10 means a worse outcome).

SECONDARY OUTCOMES:
240 Minute Pain Score | 240 minutes after enrollment.
  Self reported pain score using the Faces Pain Scale-Revised. Values range from 1-10 (10 means a worse outcome).
Oral Morphine Equivilents | From admission to the emergency department to hospital discharge, up to 72 hours.
  Opioid medications received. All opioids will be converted to oral morphine equivilents using the opioid equianalgesic calculator developed the Faculty of Pain Medicine, Australian and New Zealand College of Anesthetists (FPM ANZCA).
Parental Satisfaction | From admission to the emergency department to discharge from the emergency department, up to 72 hours.
  Participants parents/guardians will be asked to complete a satisfaction survey.
Percentage of Patients Experiencing Adverse Events | From admission to the emergency department to hospital discharge, up to 72 hours.
  Adverse events and complications will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Zachary W Binder, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (10):
- United States (9):
  - University of California, San Diego, San Diego, California
  - University of California, San Fransisco, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - UMass, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
- Gold Coast Hospital and Health Service, Southport, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data with external researchers.

REFERENCES:
- [Derived] Binder ZW, Ng C, Klekowski N, Lawson SL, Riera A, Toney AG, Pade KH, The TS, Shaahinfar A, Chaudoin LT, Lauer E, Snelling PJ, Moake MM. Ultrasound-Guided Nerve Block for Pediatric Femur Fractures in the Emergency Department: A Prospective Multi-Center Study. Acad Emerg Med. 2025 Dec;32(12):1278-1287. doi: 10.1111/acem.70084. Epub 2025 Jun 17. PMID 40524602